CLINICAL TRIAL: NCT05290168
Title: Normal Vascular Doppler Pattern of Abdominal Organ in Children
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jin-Tae Kim, Professor, Seoul National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: H2105-151-1222
Record Dates: First submitted 2022-01-17; First posted 2022-03-22 (Actual); Last update posted 2022-05-05 (Actual); Status verified 2022-05

CONDITIONS: Normal Children

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Normal children (Experimental): normal children undergoing simple surgery
  Interventions: Diagnostic Test: abdominal Doppler

INTERVENTIONS:
Diagnostic Test: abdominal Doppler — 1. Inferior vena cava diameter and distensibility
  2. Hepatic vein Doppler
  3. Portal vein Doppler
  4. Splenic artery and vein Doppler
  5. Renal artery and vein Doppler

SUMMARY:
The following ultrasonic findings are obtained at both time points before and after induction of anesthesia (T1) and after induction (T2) in normal children . Positive pressure ventilation (Tidal volume of 6-8 ml/kg and a positive exhalation pressure of 5 cmH2O) is applied after anesthetic induction.

1. Inferior vena cava diameter and distensibility
2. Hepatic vein Doppler
3. Portal vein Doppler
4. Splenic artery and vein Doppler
5. Renal artery and vein Doppler Based on this, the reference values for Doppler findings before and after anesthesia in normal children are obtained.

ELIGIBILITY:
Inclusion Criteria:

* Children undergoing simple surgery

Exclusion Criteria:

* thoracic/abdominal surgery
* surgery for congenital heart disease
* disease involving liver, kidney, spleen
* vascular disease

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-03-28 (Actual); Primary Completion 2022-12-30 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
portal vein flow velocity (cm/s) during self respiration | just before anesthesia induction (about 5 minutes before anesthetic induction)
portal vein flow velocity (cm/s) during general anesthesia | during positive pressure ventilation (within 5 - 60 minutes after anesthetic induction)
splenic vein flow velocity (cm/s) during self respiration | just before anesthesia induction (about 5 minutes before anesthetic induction)
inferior vena cava diameter (mm) during self respiration | just before anesthesia induction (about 5 minutes before anesthetic induction)
inferior vena cava diameter (mm) during general anesthesia | during positive pressure ventilation (within 5 - 60 minutes after anesthetic induction)
hepatic vein flow velocity (cm/s) during self respiration | just before anesthesia induction (about 5 minutes before anesthetic induction)
hepatic vein flow velocity (cm/s) during general anesthesia | during positive pressure ventilation (within 5 - 60 minutes after anesthetic induction)
renal artery/vein flow velocities (cm/s) during self respiration | just before anesthesia induction (about 5 minutes before anesthetic induction)
renal artery/vein flow velocities (cm/s) during general anesthesia | during positive pressure ventilation (within 5 - 60 minutes after anesthetic induction)

CONTACTS AND LOCATIONS:
Locations (1):
- Jin-Tae Kim, Seoul, South Korea